CLINICAL TRIAL: NCT06240286
Title: Comparing Manual and Neurocognitive Skills-While Sitting, Standing, Walking on a Treadmill and Using a Stepper.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Francisco Lopez-Jimenez, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-005471
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Neurocognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): Healthy subjects will attend the the Active Wellness Office at the Dan Abraham Healthy Living Center (DAHLC) at Mayo Clinic in Rochester, Minnesota, for four consecutive days. On day one, individuals will use a sitting workstation (control); based on randomization, three active workstations (standing, stepping, or walking stations) will be randomly assigned on the following days (2-4).
  Interventions: Behavioral: Sitting workstation; Behavioral: Standing workstation; Behavioral: Stepping workstation; Behavioral: Walking workstation

INTERVENTIONS:
Behavioral: Sitting workstation — Subjects will conduct reasoning, memory, concentration, and fine motor skills (neurocognitive function) assessments on a computer station in a seated position.
Behavioral: Standing workstation — Subjects will conduct reasoning, memory, concentration, and fine motor skills (neurocognitive function) assessments on a computer station while standing.
Behavioral: Stepping workstation — Subjects will conduct reasoning, memory, concentration, and fine motor skills (neurocognitive function) assessments on a computer station while utilizing a stepper.
Behavioral: Walking workstation — Subjects will conduct reasoning, memory, concentration, and fine motor skills (neurocognitive function) assessments on a computer station while walking on a treadmill.

SUMMARY:
This study is being performed to evaluate the effect of different active workstations (e.g., standing, stepping, or walking stations) on work performance through the evaluation of neurocognitive function using reasoning, memory, concentration, and fine motor skills evaluation tools.

ELIGIBILITY:
Inclusion Criteria:

* Dan Abraham Healthy Living Center (DAHLC) members and non-members that have provided informed consent to participate in this study.

Exclusion Criteria:

* Unable to stand up, walk on a treadmill or use a stepper.
* Alzheimer, dementia or any memory impairment.
* Cannot attempt fine motor skills.
* Not willing to use a treadmill, stepper or standing desk.
* Not a present user of an active office.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Double Trouble Task Score | Day 1, Day 2, Day 3, Day 4
  The Double Trouble Task is a computer based reasoning assessment that evaluates the Stroop effect which relates to the increased difficulty a person has in naming the print color of a word when the text of that word refers to an 'incongruent' color. It evaluates the capacity to inhibit automatic word recognition by selectively focusing the attention to impede the automated access of distracting word information. In the website version, three words appear on the screen, one at the top, and two at the bottom. Subjects click the word at the bottom that matches the color at the top for 90 seconds and 1 point for each correct answer. Higher scores represent better reasoning skills & neurocognitive function.
Grammatical Reasoning Test Score | Day 1, Day 2, Day 3, Day 4
  The Grammatical Reasoning Test is a computer based reasoning assessment that measures the capacity of a person to reason the relationships among different objects and shapes. A statement appears at the top of the screen with two shapes at the bottom. Participants clicked on 'True' or 'False' to indicate whether the sentence accurately described the relationship between the shapes in 90 seconds and participants obtained 1 point for each correct answer. Higher scores represent better reasoning skills & neurocognitive function.
Odd One Out Test Score | Day 1, Day 2, Day 3, Day 4
  The Odd One Out Test is a computer based reasoning assessment which evaluates the person's Intelligence Quotient. It measures fluid intelligence or the capacity to reason abstractly and solve problems. Derived from Raven's and Cattell's intelligence tests. During the test, 9 patterns (color, shape, and number) appeared on the screen; participants chose the pattern (odd one) that differed from the others for 3 minutes and got 1 point for each correct answer. Higher scores represent better reasoning skills & neurocognitive function.
Object Reasoning Task Score | Day 1, Day 2, Day 3, Day 4
  The Object Reasoning Task is a computer based reasoning assessment that evaluates an individual's capability to make logical deductions from a sequence of complex images. Subjects look at 4 panels, 3 at the top and 1 at the bottom. Each panel contained four separate diagrams; subjects decided whether the panel at the bottom was the next in the series or not. It takes 3 minutes and 1 point for each correct answer. Higher scores represent better reasoning skills & neurocognitive function.
Spatial Span Task Score | Day 1, Day 2, Day 3, Day 4
  The Spatial Span Task is a computer based memory assessment that assesses the visuospatial working memory that depends on the unitary short-term memory system. Participants must remember a sequence of flashing boxes and click to the correct order; when they make a mistake the test ends and they have 3 opportunities. When they click in the right order, the following sequence increases difficulty. 4 points are the baseline; for each correct answer subjects get 1 point; if incorrect, they lose points. Higher scores represent better memory skills & neurocognitive function.
Monkey Ladder Task Score | Day 1, Day 2, Day 3, Day 4
  The Monkey Ladder Task is a computer based memory assessment that assesses the visual working memory better developed in chimpanzees than humans. Participants must remember which number appears in specific boxes, after a short period, the numbers disappear and they have to click on the boxes in numerical sequence, after three errors the test ends. 2 points are the baseline. Participants get 1 point for the correct answers; if incorrect, they lose the points earned. Higher scores represent better memory skills & neurocognitive function.
Digit Span Task Score | Day 1, Day 2, Day 3, Day 4
  The Digit Span Task is a computer based memory assessment that evaluates the verbal working memory that allows the temporary storage and manipulation of information. Participants must remember a sequence of numbers by typing them using the keyboard; after typing the correct sequence of numbers, the difficulty increases and after 3 mistakes the test ends. Participants get 1 point for a proper sequence; if incorrect, they lose points. Higher scores represent better memory skills & neurocognitive function.
Paired Associates Task Score | Day 1, Day 2, Day 3, Day 4
  The Paired Associates Task is a computer based memory assessment that assesses the paired-associate learning skills, a mental skill that requires learning to pair two items in memory. When the difficulty increases, several regions in the brain activate. During the task, a set of boxes appear on the screen. The boxes open, one after the other to reveal the figure inside, and subjects must remember and click which figure appears in which box. The difficulty increases in the number of figures after clicking the correct sequence and subjects will have three opportunities. Participants get 1 point for the right answers; if incorrect, they lose the points. Higher scores represent better memory skills & neurocognitive function.
Rotations Task Score | Day 1, Day 2, Day 3, Day 4
  The Rotations Task is a computer based concentration assessment that measures the ability to rotate objects mentally. Two rotated boxes appear on the screen, each filled with red and green squares. Participants click the boxes 'Match' or 'Mismatch' in 90 seconds, if the answer is correct, they get 8 points; if not, they lose the points. Higher scores represent better concentration skills & neurocognitive function.
Feature Match Task Score | Day 1, Day 2, Day 3, Day 4
  The Feature Match Task is a computer based concentration assessment that measures perception, requires concentration and focuses on complex images. Two boxes appear on the screen one at the left and the other to the right, each containing a complex array of abstract shapes. Subjects will click if the figures 'Match' or 'Mismatch' for 90 seconds. If correct, the next problem will be more difficult. The points are given according to the problem's difficulty; they can vary from 1-11and above. Higher scores represent better concentration skills & neurocognitive function.
Polygons Task Score | Day 1, Day 2, Day 3, Day 4
  The Polygons Task Score is a computer based concentration assessment that measures the mental ability to compare complex images. Two overlapping images appear on one side of the monitor, and another figure appears on the other side and contains just one shape. Subjects click 'Match' or 'Mismatch' to indicate if the single figure is identical or different in shape from one of the overlapping figures. Each chance will increase in difficulty. Subjects in 90 seconds will try to score as many points as they can, points per correct answer can vary from 1-6 points and above. Higher scores represent better concentration skills & neurocognitive function.
Typing Test Score | Day 1, Day 2, Day 3, Day 4
  The Typing Test is a computer based fine motor skills assessment. It is measured using the Split Screen Typing Program (Typing Master Inc., Helsinki, Finland). Subjects completed a 3-minute test typing as fast and accurately as they could, the top of the screen showed the text that participants had to type, and the typed text was seen at the bottom of the computer monitor. Participants typed one different script for each station. Typing speed, as well as accuracy represented by number of errors, and adjusted individual typing speed at each workstation were scored. The higher typing speed & accuracy scores (low number of errors) represent better fine motor skills.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lopez-Jimenez, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medina-Inojosa JR, Gomez Ibarra MA, Medina-Inojosa BJ, Supervia M, Jenkins S, Johnson L, Suarez NP, Bonikowske A, Somers VK, Lopez-Jimenez F. Effect of Active Workstations on Neurocognitive Performance and Typing Skills: A Randomized Clinical Trial. J Am Heart Assoc. 2024 Apr 16;13(8):e031228. doi: 10.1161/JAHA.123.031228. Epub 2024 Apr 4. PMID 38572691